CLINICAL TRIAL: NCT02047760
Title: Investigation Into the Role of Neuroretinal Biomarkers in the Phenotyping of Neurodegenerative Diseases, and Potential for Tracking Progression and Monitoring Impact of Interventions, Events and Therapies.
Brief Title: Neuroretinal Biomarkers in Neurodegenerative Diseases
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 147305
Record Dates: First submitted 2014-01-22; First posted 2014-01-28 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MS patients: All MS sub-types
- Controls: sex- and age-matched controls

SUMMARY:
There is increasing evidence that examining our eyes can tell us a lot of information about our health, and systemic diseases. We want to study what eyes can reveal about serious neurodegenerative diseases like multiple sclerosis, and motor neurone disease, by analysing the retinal images from a simple non-invasive eye scan, that is already being routinely used to provide immediate clinical information in this group of patients.

DETAILED DESCRIPTION:
The identification of reliable biomarkers in multiple sclerosis (MS), and other neurodegenerative diseases, has become increasingly important with the development of disease-modifying treatments.

A range of genetic, metabolic and imaging biomarkers exist, in correlations with diagnosis, phenotypic expression, inflammation, degeneration and prognosis; although there is wide variation in specificity, sensitivity, reproducibility and cost.

In MS specifically, we know that whilst the primary pathological process is demyelination of neurones (which can be accompanied by inflammation, and resolving symptoms), it is the subsequent axonal loss - neurodegeneration - that gives rise to the permanent functional disability.

Magnetic resonance imaging (MRI) brain scans are currently our primary source of objective information in assessing MS disease status, in terms of neurodegeneration and possibly prognosis. Measurements of brain atrophy have shown worsening rates are higher in untreated MS patients compared with healthy controls and also correlate with subsequent disability status eight years later.

However, brain atrophy measures sometimes reveal paradoxical outcomes, particularly of white matter atrophy, where normal or increased volume as a result of pathological processes, such as tissue damage and repair, can impact upon the measures.

The search then for other markers of neurodegenerative disease status and prognosis continues, with renewed interest in the eye.

In MS, early work has suggested certain retinal measures, particularly the width of the layer that consists largely of retinal ganglion cell nerve axons, as candidate biomarkers, under the hypothesis that neuroretinal tissue reflects global central nervous system (CNS) pathology. Conceptually, this would seem reasonable, given the frequency for anterior visual pathway involvement as the primary presentation of MS; and in addition, the unmyelinated ganglion cell axons that form the retinal nerve fibre layer (RNFL) are a direct extension of the brain, and global neurodegeneration would be expected to involve these neurones - particularly in MS, where the disease lesions have a predilection for the periventricular regions, which are in close proximity to the optic radiations.

However, the natural history of neuroretinal tissue integrity is poorly understood, and in vivo measurement is a very new modality, requiring validation and context to any interpretation.

In addition, retinal imaging permits the direct visualisation, and subsequent analysis, of the retinal vasculature - shown in studies of stroke and hypertension to be an accurate representation of brain vasculature, with diagnostic and prognostic potential.

In summary, a combined score of neuroretinal integrity as measured by retinal imaging may yield new insights into sever neurodegenerative disease.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate with informed consent
* age 18-75
* male or female
* confirmed diagnosis of multiple sclerosis

Exclusion Criteria:

* concurrent eye disease, or media opacity
* high refractive error (> +6 or -6)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All MS patients attending the ARRNC research clinic
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Retinal nerve fibre layer (RNFL) thickness change over time | 0, 6, 12, 24 months
  Monitoring of RNFL thickness over time, as measured by optical coherence tomography (OCT) retinal scanning, particularly in relation to disease events, or interventions.

SECONDARY OUTCOMES:
Retinal vascular fractal dimension change over time | 0, 6, 12, 24 months
  Monitoring of retinal vessel metrics, of bifurcation optimality and tortuosity; and combination with neuroretinal measures as a combined score.

CONTACTS AND LOCATIONS:
Overall Officials: James Cameron, FRCOphth, Principal Investigator — University of Edinburgh
Locations (1):
- Anne Rowling Regenerative Neurology Clinic, Edinburgh, United Kingdom